CLINICAL TRIAL: NCT02322671
Title: An Open-label, Randomised, Single Dose, Three-Way Crossover, Six Sequence, Pilot Study to Determine the Relative Bioavailability of Montelukast Sodium 5mg From Two Candidate Chewable Tablet Formulations of GW483100 Relative to One 5mg Chewable Tablet of Reference Montelukast Sodium in Healthy Adult Subjects Under Fasting Conditions
Brief Title: Relative Bioavailability Study of Two Montelukast Sodium (GW483100) 5 Milligrams (mg) Chewable Tablets and One Reference Montelukast Sodium 5 mg Chewable Tablet in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200107
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Disorders
Keywords: chewable tablet; montelukast sodium; healthy adult subjects; relative bioavailability; GW483100
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence ABC (Experimental): Subjects will be administered a single oral dose of treatment A, B and C in the sequence ABC, where A is Reference Treatment: 5 mg montelukast sodium reference chewable tablets (innovator product); B is Test Formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and C is Test Formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days
  Interventions: Drug: Reference Montelukast; Drug: Test 1 Montelukast; Drug: Test 2 Montelukast
- Sequence ACB (Experimental): Subjects will be administered a single oral dose of treatment A, B and C in the sequence ACB, where A is Reference Treatment: 5 mg montelukast sodium reference chewable tablets (innovator product); B is Test Formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and C is Test Formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days
  Interventions: Drug: Reference Montelukast; Drug: Test 1 Montelukast; Drug: Test 2 Montelukast
- Sequence BAC (Experimental): Subjects will be administered a single oral dose of treatment A, B and C in the sequence BAC, where A is Reference Treatment: 5 mg montelukast sodium reference chewable tablets (innovator product); B is Test Formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and C is Test Formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days
  Interventions: Drug: Reference Montelukast; Drug: Test 1 Montelukast; Drug: Test 2 Montelukast
- Sequence BCA (Experimental): Subjects will be administered a single oral dose of treatment A, B and C in the sequence BCA, where A is Reference Treatment: 5 mg montelukast sodium reference chewable tablets (innovator product); B is Test Formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and C is Test Formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days
  Interventions: Drug: Reference Montelukast; Drug: Test 1 Montelukast; Drug: Test 2 Montelukast
- Sequence CAB (Experimental): Subjects will be administered a single oral dose of treatment A, B and C in the sequence CAB, where A is Reference Treatment: 5 mg montelukast sodium reference chewable tablets (innovator product); B is Test Formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and C is Test Formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days
  Interventions: Drug: Reference Montelukast; Drug: Test 1 Montelukast; Drug: Test 2 Montelukast
- Sequence CBA (Experimental): Subjects will be administered a single oral dose of treatment A, B and C in the sequence CBA, where A is Reference Treatment: 5 mg montelukast sodium reference chewable tablets (innovator product); B is Test Formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and C is Test Formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days
  Interventions: Drug: Reference Montelukast; Drug: Test 1 Montelukast; Drug: Test 2 Montelukast

INTERVENTIONS:
Drug: Reference Montelukast — It is available as pink, round, bi-convex-shaped chewable tablet of reference 5 mg montelukast sodium (innovator product). that has to be placed on the tongue and chewed immediately.
Drug: Test 1 Montelukast — It will be provided as pink, round, bi-convex-shaped chewable tablet of test formulation 1: 5mg montelukast sodium (GW483100) that has to be placed on the tongue and chewed immediately.
Drug: Test 2 Montelukast — It will be provided as pink, round, bi-convex-shaped chewable tablet of test formulation 2: 5mg montelukast sodium (GW483100) that has to be placed on the tongue and chewed immediately.

SUMMARY:
This study is designed to estimate the bioavailability of montelukast from the 5 milligrams (mg) montelukast sodium (GW483100) test formulations relative to 5 mg montelukast sodium reference chewable tablets (innovator product). It is an open-label, randomized, single dose, three-way cross over, six sequence study in 18 healthy human subjects. Each subject will participate in all three treatment periods. Subjects will be randomized to one of six sequences and administered one of the three treatments A, B or C in each treatment period, where Treatment A is 5mg chewable tablet of reference 5 mg montelukast sodium reference chewable tablets (innovator product), Treatment B is test formulation 1: 5mg montelukast sodium (GW483100) chewable tablet and Treatment C is test formulation 2: 5mg montelukast sodium (GW483100) chewable tablet. The treatment periods will be separated by a washout period of 7 to 14 days. Total duration in the study for each subject will be approximately 8 weeks from screening to the follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Male and females aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required, agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilograms (kg) and Body mass index (BMI) within the range 19 - 24.9 kilograms per square meter (kg/m^2) (inclusive).
* Male subject
* Female subject: is eligible to participate if she is not pregnant (as confirmed by a negative serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

Non-reproductive potential defined as:

Pre-menopausal females with one of the following:

Documented tubal ligation Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion Hysterectomy Documented Bilateral Oophorectomy

* Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until [at least five terminal half-lives OR until any continuing pharmacologic effect has ended, whichever is longer] after the last dose of study medication and completion of the follow-up visit.

GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP This list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis.

* Contraceptive subdermal implant that meets the standard operating procedure (SOP)effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches
* Male partner sterilisation with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository) only for the following 3 situations when there is a very low risk for developmental toxicity: Vaccines; Monoclonal antibodies when there is no target biology concern; Compounds that have a complete reproductive toxicology package and have not shown any signal for developmental toxicity.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.

* Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until [at least five half-lives of study medication or for a cycle of spermatogenesis following five terminal half-lives] after the last dose of study medication.
* Vasectomy with documentation of azoospermia.
* Male condom plus partner use of one of the contraceptive options below:
* Contraceptive subdermal implant that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Oral Contraceptive, either combined or progestogen alone. Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and bilirubin >1.5 x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Corrected QT (QTC) > 450 milliseconds (msec)
* NOTES: The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machineread or manually over-read.
* The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.
* For purposes of data analysis, QTcB, QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).
* No concomitant medications should be taken by the subject while participating in the study. Refer to Study Protocol for further detail.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Subjects with phenylketonuria
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment. For potent immunosuppressive agents, subjects with presence of hepatitis B core
* A positive pre-study drug/alcohol screen.
* A positive test for Human Immunodeficiency Virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* Any symptoms with a systolic Blood pressure (BP) <95 millimeters of mercury (mmHg)
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing
* Lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2015-04-20 (Actual); Study Completion 2015-04-20 (Actual)

PRIMARY OUTCOMES:
Composite of plasma pharmacokinetic [PK] parameters of montelukast sodium | Pre-dose, 0.50, 1.00, 1.25, 1.50, 1.75, 2.0, 2.25, 2.50, 2.75, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post dose during each treatment period
  Plasma PK parameters includes Maximum observed concentration (Cmax), Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite[inf] time (AUC[0-inf]) and Area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration within a subject across all treatments (AUC[0-t]).

SECONDARY OUTCOMES:
Composite of plasma PK parameters of montelukast sodium | Pre-dose, 0.50, 1.00, 1.25, 1.50, 1.75, 2.0, 2.25, 2.50, 2.75, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 16.00 and 24.00 hours post dose during each treatment period
  Plasma PK parameters includes time of occurrence of Cmax (tmax), Percentage of AUC(0-inf) obtained by extrapolation (%AUCex) and Terminal phase half-life (t½)
Number of subjects with Adverse Events (AEs) | Up to 8 weeks
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.
Blood pressure assessments | Up to 5 weeks
  In each treatment period, systolic and diastolic blood pressure will be measured in supine position after 5 minutes(min) rest at pre-dose (-2.00 to 0.00 hours.), 1, 2, 4, 8, 12 and 24 hours within ±30min.
Pulse rate assessments | Up to5 weeks
  In each treatment period, pulse rate will be measured in supine position after 5 min rest at pre-dose (-2.00 to 0.00 hours.), 1, 2, 4, 8, 12 and 24 hours within ±30min.
Clinical laboratory assessments | Day -1 and end of treatment period 3 (approximately Week 5)
  Clinical laboratory parameters includes haematology, clinical chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hyderabad, India

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200107 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200107?search=study&search_terms=200107#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200107 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register